CLINICAL TRIAL: NCT00607191
Title: Clubfoot DNA Repository
Status: Completed | Type: Observational
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Jonathan Rios, PhD, Staff Scientist, Texas Scottish Rite Hospital for Children
Other Study IDs: UTSW 122007-004
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Clubfoot
Keywords: Idiopathic talipes equinovarus (ITEV)
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each of the study participants (affected and non-affected individuals) will be asked to provide DNA from a blood sample. A 10cc sample of blood will be removed on 1 or 2 occasions by drawing blood from the arm or by finger stick by research staff. If the participant is a child who will be undergoing surgery, the blood sample will be collected at that time to eliminate additional stick. If collecting a blood sample is not possible we can also obtain DNA by collecting a saliva sample. This second technique does not give us as much DNA as we would get from blood. Therefore, if we get saliva samples, we might require more than one saliva sample over the course of the study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To build a DNA repository to enable participation in ongoing and future Clubfoot genetic linkage studies.

DETAILED DESCRIPTION:
Clubfoot is a birth defect that can occur alone (in isolation) or as a part of a disease like cerebral palsy (CP). Genetic linkage is a research tool in which DNA samples are tested for genetic landmarks (markers) whose location on chromosomes is known. Genes and markers that are physically close to one another on the chromosome are said to be tightly linked than genes and markers that are located far apart. This gives clues of where to search for genes causing isolated clubfoot. If there appears to be a high correlation between family members' inheritance of a particular marker, and their inheritance of the trait being studied (in this case clubfoot), the area of the chromosome near that marker can then be searched for a likely gene which causes the trait. It is hoped that genetic linkage research might eventually result in new or improved ways to determine individuals and families at higher risk for clubfoot and development of new or improved ways to treat clubfoot.

Our research staff will obtain information about each subject and their family called a pedigree. We will then administer a one page questionnaire to the mother(s) of the affected individual(s). This questionnaire will ask about the mother's experiences during pregnancy (e.g. Did she take multivitamins? Did she smoke or drink? etc.)

Each of the study participants (affected and non-affected individuals) will be asked to provide DNA from a blood sample. If collecting a blood sample is not possible we can also obtain DNA by collecting a saliva sample.

Samples for DNA processing will be stored according to the following repository guidelines. Patient/donor-subject information, questionnaires, and consents will be maintained by the orthopaedic research coordinator.

Samples will be made to investigators not affiliated with UT Southwestern who wish to study genetic factors that cause clubfoot; for example, we have recently been approached by Jacqueline Hecht (UT Health Science Center, Houston) and Matthew Dobbs (Washington University, St. Louis) regarding participation in their multicenter trials. Samples will be de-identified and will include no personal information which would link the sample to the donor subject.

Primary investigator and sub-investigators will determine how samples will be used and by whom. Additional research utilizing subjects' samples will be approved by the Texas Scottish Rite Hospital for Children Research Advisory Panel and the Institutional Review Board at UT Southwestern.

ELIGIBILITY:
Inclusion Criteria:

* For a family to be included in this study there should be at least one person in the family affected with Idiopathic Talipes Equinovarus (or clubfoot). If the person satisfies this criterion, then the affected person and his/her parents are included in the study. If there are other individuals in the family who are also affected (e.g. a cousin), then these individuals are also invited to participate in the study along with their parents, siblings and all other family members that link the two affected individuals (e.g. grandparents).

Exclusion Criteria:

* Inability to speak and read English or Spanish
* Should not have any other major birth defect (e.g. Heart defects, Downs Syndrome or cerebral palsy).

Ages: 1 Week to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients being treated at the participating facilities with a diagnosis of clubfoot, and their affected family members.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2008-01; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

PRIMARY OUTCOMES:
To identify a gene, or genes, that are associated with isolated clubfoot. | 10 years

SECONDARY OUTCOMES:
New or improved ways to determine individuals and families at higher risk for clubfoot and development of new or improved ways to treat clubfoot. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rios, PhD, Principal Investigator — Texas Scottish Rite Hospital for Children
Locations (1):
- Texas Scottish Rite Hospital for Children, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Texas Scottish Rite Hospital for Children — http://www.tsrhc.org